CLINICAL TRIAL: NCT02184494
Title: Phase 1 Study of A Double-Blind Placebo-Controlled Study of the Effect of Beta-Alanine and Whole Body Vibration on Neurologic Motoric Function, Vascular Function, and Quality of Life in Parkinson's Disease
Brief Title: Blood Lactate Concentrations With and Without Exercise in Parkinson's Disease and Multiple Sclerosis Patients
Acronym: PDMSLac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014:12658; HPN (Other: FSU Human Performance and Sports Nutrition)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease; Multiple Sclerosis
Keywords: Parkinson's Disease; Multiple Sclerosis; Fatigue; Resting Energy Expenditure; Whole Body Vibration; Exercise; Blood Lactate
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blood Lactate Response in PD (Experimental): This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in a PD population. One set of the squats will be performed on a whole body vibration plate (pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)), and one on the ground.
  Interventions: Device: pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)
- Blood Lactate Response in MS (Experimental): This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in an MS population. One set of the squats will be performed on a whole body vibration plate (pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)), and one on the ground.
  Interventions: Device: pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)
- Blood Lactate Responses in Controls (Experimental): This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in healthy, older adults. One set of the squats will be performed on a whole body vibration plate (pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)), and one on the ground.
  Interventions: Device: pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands)

INTERVENTIONS:
Device: pro5 AIRdaptive Power Plate (Badhoevedorp, The Netherlands) — Subjects will be exposed to vertical vibration with a frequency and peak-to-peak displacement of 30 Hz and 1 mm, respectively, which provides a peak-to-peak acceleration of about 4.16 G.
  Whole Body Vibration

SUMMARY:
Fatigue is one of the most common and debilitating symptoms experienced in Parkinson's Disease (PD) and Multiple Sclerosis (MS). There are multiple proposed mechanisms of disorder-related fatigue, however, it is unknown whether PD or MS patients experience compromised blood lactate responses to an acute bout of exercise, subjecting them to exercise-related fatigue. These populations may experience higher energy expenditure at rest due to increased rigidity, however, limited data exists investigating resting energy expenditure in these populations.

Researchers hypothesize that PD and MS patients will display higher resting energy expenditure than healthy age-matched controls, and that level of energy expenditure will correlate with amount of rigidity or spasticity. Also, we hypothesize that baseline levels of lactate will not be different between PD/MS and control groups, but post-exercise blood lactate levels will be significantly higher in the PD/MS groups.

DETAILED DESCRIPTION:
Patients diagnosed with Parkinson's Disease (PD) and Multiple Sclerosis (MS) frequently experience increased levels of muscle weakness and fatigue; This impairment is exacerbated with onset of exercise and alleviated with rest or sleep . Importantly, in about 1/3 of PD patients, fatigue is considered debilitating , and even further, there is inconclusive evidence suggesting that anti-PD and anti-MS drugs improve fatigue. The precise mechanisms and pathogenesis of the disorder-specific fatigue in PD and MS remain elusive.

Both peripheral and central cholinergic systems are affected in PD , however, it has been shown that peripheral cholinergic neurons at the neuromuscular junction are normal functioning . Even so, recruitment of necessary motor units may be greatly affected due to peripheral neuropathy common in both PD and MS . Following repetitive nerve stimulation in PD and MS, there is consistent evidence of a decrease in the number of functioning motor units and decrements in muscle responses. This promotes progressive fatigue with decrements in the amplitude of movement. Therefore, recruitment of motor units may be a major cause of rapid fatigue in repetitive movement with PD and MS patients, even though peripheral neuromuscular junctions do not seem to be affected. In addition to skeletal muscle inefficiency, work rate and efficiency of breathing using respiratory muscles is significantly lower in a PD population during repetitive stimulation, used to simulate exercise-induced repetitive contractions. Respiratory inefficiencies in MS include, but are not limited to reduced forced vital capacity, hypoxemia, and respiratory muscle weakness.

In addition to possible neurological mechanisms of PD- and MS-related fatigue, rigidity, defined as involuntary state of continuous muscle tension in PD, and spasticity and rigidity in MS may also have a profound effect on fatigue outcomes . Adequate muscle length is required for effective muscle contraction. Rigidity likely changes the length of the muscle at rest, and therefore contributes to ineffective muscle contraction when active. In addition to inefficient muscle contraction, the increased continuous active contraction, or tone, of the muscle results in an increase in resting energy expenditure compared to healthy individuals, even in pharmacologically treated PD patients. Interestingly, resting energy expenditure in MS patients was shown to be comparable to age-matched healthy controls; however, it is important to note that these MS patients remained medicated during the study. In addition, rigidity and spasticity, common in PD and MS, respectively may provide varying levels of resting energy expenditure; however, no research to date has examined these differences. In total, if more energy is being expended at rest, hypothetically, PD and MS patients will have inadequate energy stores to exercise to their respective full capacity. This could potentiate early onset of lactic acid and hydrogen accumulation in active muscle, decrease the pH of the active muscle, and contribute to early fatigue in repetitive tasks.

Purportedly, the combination of early onset of skeletal and respiratory muscle fatigue, in addition to muscle rigidity would create an environment similar to that of high intensity exercise, even at low intensities or rest. The ensuing result may likely be an accumulation of lactic acid and hydrogen ions, making the muscle environment very acidic. However, changes in the levels of resting and post-exercise blood lactate levels have not been elucidated. Therefore, we are planning to measure resting energy expenditure using a ventilation face mask and a noseclip. Blood lactate will be sampled at rest, after simulated high-intensity exercise, and ten minutes after rest (when lactate significantly increases). The exercise will consist of performing 5 sets of static, shallow 120 degree squats for 1 minute, with 1 minute of seated rest between each squat. Sustained isometric contraction at 2/3 of the maximal voluntary contractile force for 2 to 3 minutes was found to occlude local blood flow enough that local oxygen stores were depleted . Muscle lactate is also increased 12-fold upon fatigue of isometric holds such as squats. This same environment of lactic acid buildup can be simulated by circulatory occlusion as well as 60-second isometric quadricep contractions . Isometric squats will be employed to observe differences in blood response in PD compared to healthy individuals.

Therefore, the purpose of this study is to analyze the differences in resting energy expenditure and exercise-induced lactate production in PD and MS compared to healthy, age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease Stage I-IV (be standard criteria H&Y scale)
* Multiple Sclerosis
* Healthy, age-matched controls
* 45 to 90 years old

Exclusion Criteria:

* Dementia
* Co-morbid neurologic factors
* Individuals without independent ambulation
* Significant heart and respiratory disease
* Debilitating arthritis

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ormsbee, Ph.D., Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Fitness and Wellness Center, Tallahassee, Florida
  - Balance Disorders Clinic, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Yes
If, and when requested, participants may review findings by contacting the PI. Other than participants, only investigators will have access to the data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Lactate Response in PD: This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in a PD population. One set of the squats will be performed on a whole body vibration plate, and one on the ground.
  pro5 AIRdaptive Power Plate, Badhoevedorp, The Netherlands: Subjects will be exposed to vertical vibration with a frequency and peak-to-peak displacement of 30 Hz and 1 mm, respectively, which provides a peak-to-peak acceleration of about 4.16 G.
  Whole Body Vibration
- Blood Lactate Response in MS: This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in an MS population. One set of the squats will be performed on a whole body vibration plate, and one on the ground.
  pro5 AIRdaptive Power Plate, Badhoevedorp, The Netherlands: Subjects will be exposed to vertical vibration with a frequency and peak-to-peak displacement of 30 Hz and 1 mm, respectively, which provides a peak-to-peak acceleration of about 4.16 G.
  Whole Body Vibration
- Blood Lactate Responses in Healthy, Older Adults: This arm involves performing 5 sets of 1-minute squats with 1 minute of rest between each, and a finger prick before, after, and 10 minutes after the exercise in healthy, older adults. One set of the squats will be performed on a whole body vibration plate, and one on the ground.
  pro5 AIRdaptive Power Plate, Badhoevedorp, The Netherlands: Subjects will be exposed to vertical vibration with a frequency and peak-to-peak displacement of 30 Hz and 1 mm, respectively, which provides a peak-to-peak acceleration of about 4.16 G.
  Whole Body Vibration
Period: Overall Study
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Started | 13 | 13 | 8
Completed | 12 | 11 | 8
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults | Total
Number analyzed (Participants) | 12 | 11 | 8 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 7 | 19
  >=65 years | 9 | 2 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9) | 52 (10) | 50 (10) | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 7 | 25
  Male | 5 | 0 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Blood Lactate Response
Description: Measured using a blood lactate analyzer, a finger prick test measured before, after, and 10 minutes after exercise
Time Frame: Before, immediately after, and 10 minutes after the squatting exercise protocol
Population: 2 of the 8 participants in the healthy, older adults group did not return for this visit, and thus, were not included in analysis.
  1 of the 12 MS participants did not return for this visit, and thus, were not included in analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Number analyzed (Participants) | 12 | 11 | 6
mmol/L
  Pre without Whole Body Vibration | 1.7 (0.7) | 1.6 (0.7) | 1.2 (0.4)
  Immediately Post without Whole Body Vibration | 2.3 (0.9) | 2.8 (1.3) | 2.5 (1.1)
  10 Minutes Post without Whole Body Vibration | 2.2 (1.3) | 3.3 (2.3) | 2.6 (1.2)
  Pre with Whole Body Vibration | 1.8 (0.7) | 2.2 (1.0) | 1.3 (0.3)
  Immediately Post with Whole Body Vibration | 3.1 (2.4) | 4.3 (3.0) | 2.9 (0.9)
  10 Minutes Post with Whole Body Vibration | 1.8 (0.5) | 3.1 (1.9) | 2.2 (0.9)

2. Secondary Outcome: Resting Energy Expenditure
Description: Measured using using indirect calorimetry with a ventilated face mask and noseclip (Parvometrics, Sandy, UT). This involves laying supine for 30 to 60 minutes.
Time Frame: Measured immediately upon arriving to the laboratory. Lasted approximately 25 minutes.
Population: 1 of the 12 PD participants had severe claustrophobia, and could not tolerate the breathing mask on their face.
  1 of the 12 PD participants, and 1 of the 8 healthy, older adults participants: dysfunctional equipment, and thus invalid results.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Number analyzed (Participants) | 10 | 11 | 7
kcal | 1338 (284) | 1262 (139) | 1521 (276)

3. Other Pre Specified Outcome: Neurological Function
Description: Neurological functional state will be assessed using the Unified Parkinson's Disease Rating Scale (UPDRS). Of the 5 sections of the examination, two parts were used. Part II (self-evaluation of aspects of the experiences of daily living) consisted of 13 Likert scale questions (graded 0 to 4, with 4 being most severe), including speech, saliva and drooling, chewing and swallowing, eating tasks, dressing, hygiene, handwriting, doing hobbies and other activities, turning in bed, tremor, getting out of bed/car/deep chair, walking and balance, and freezing. Part III (motor evaluation performed by trained research personnel) consisted of 14 Likert scale questions (graded 0 to 4, with 4 being most severe), including speech, facial expression, rigidity, finger tapping, hand movements, pronation-supination movements of hands, toe tapping, leg agility, arising from chair, gait, etc... Values were summed, with higher values indicating increased impairment and disability.
Time Frame: Measured immediately after the resting energy expenditure measurement, and before the other questionnaires. Lasted approximately 15 minutes.
Population: The MS and healthy, older adults populations were not required to be assessed with the UPDRS because the assessment materials were for PD populations, specifically.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Number analyzed (Participants) | 12 | 0 | 0
units on a scale | 23 (6) |  |

4. Other Pre Specified Outcome: Health and Activity Questionnaire
Description: Short Form 36 Health Survey questionnaire: patient-reported survey of 36 questions, yielding the participant's degree of health on 8 different scale scores (each scale summed into a 0-100 score, with lower scores indicating more disability). The eight scales include vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.
  Schwab and England Activities of Daily Living Questionnaire: self-rated, single item assessment of the participant's ability to perform daily activities with speed and independence, measured using a Likert scale of percentages, in 10% increments. A score of 100% indicates total independence, while 0% indicates complete dependence.
Time Frame: Collected immediately after the UPDRS (if PD population), or immediately after the resting energy expenditure measurement (if MS or healthy, older adult). Measured with other questionnaires and immediately before squatting exercise. Lasted ~10 minutes.
Population: 2 of the 8 healthy, older adults did not complete all of the surveys, and were thus, clearly unable to be added to analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Number analyzed (Participants) | 12 | 11 | 6
units on a scale
  Physical Funcitoning | 65 (21) | 66 (22) | 95 (4)
  Role Limitations due to Physical Health | 43 (34) | 70 (32) | 82 (35)
  Role Limitations due to Emotional Health | 73 (34) | 82 (26) | 90 (23)
  Energy/Fatigue | 55 (17) | 42 (26) | 71 (21)
  Emotional Well-Being | 75 (16) | 75 (13) | 87 (5)
  Social Functioning | 78 (20) | 73 (22) | 95 (13)
  Pain | 73 (16) | 70 (29) | 86 (8)
  General Health | 68 (19) | 58 (15) | 87 (8)
  Activities of Daily Living | 85 (5) | NA (NA) — Participants in this group did not complete this survey. | 100 (0)

5. Other Pre Specified Outcome: Fatigue/Depression Assessment
Description: Fatigue Severity Scale: 9-item, self-reporting rating that rates the severity of your fatigue symptoms on a Likert scale ranging from 1 to 7, with 1 indicating strong disagreement, and 7 indicating strong agreement. The sum of scores is calculated. The lower the score, the more severe the participant's fatigue symptoms.
  Beck's Depression Inventory: 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression on a Likert scale ranging from 0 to 3, with 3 being the most severe. The sum of scores is calculated. A high score indicates more severe depression and related symptoms.
Time Frame: Collected at the same time as the other questionnaires. Lasted approximately 5-7 minutes.
Population: 2 of the 8 healthy, older adults did not complete all of the surveys, and were thus unable to be added to analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Number analyzed (Participants) | 12 | 11 | 6
units on a scale
  Depression | 7 (5) | 8 (5) | 3 (3)
  Fatigue | 30 (18) | 38 (17) | 17 (14)

ADVERSE EVENTS:
Time Frame: During the study collection period
Description: Subjects were asked about any adverse affects.
Arm/Group | Blood Lactate Response in PD | Blood Lactate Response in MS | Blood Lactate Responses in Healthy, Older Adults
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes